CLINICAL TRIAL: NCT01338961
Title: Normothermia Versus Hypothermia for Patients With Valvular Heart Disease Operated Under Cardiopulmonary Bypass.
Brief Title: Normothermia Versus Hypothermia for Valvular Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Efremov Sergey, Anesthesist, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HYPO-2010
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Valvular Heart Disease
Keywords: Cardiopulmonary Bypass; Hypothermia; Normothermia; Troponin I; Bleeding
MeSH Terms: conditions — Heart Valve Diseases; Hypothermia; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normothermic CPB (No Intervention): Standard management. Patients will be kept at normothermia throughout the procedure (>36oC).
- Hypothermic CPB (Active Comparator): Patients will be cooled to 31-32oC (nasopharyngeal) after the beginning of CPB. Rewarming will begin 10-15 min before release of aortic cross-clamp. The gradient between heat-exchanger and nasopharynx during rewarming will be maintained at 3oC. The rewarming will be stopped at 36,5oC.
  Interventions: Procedure: Hypothermic CPB

INTERVENTIONS:
Procedure: Hypothermic CPB — Patients will be cooled to 31-32oC (nasopharyngeal) after the beginning of CPB. Rewarming will begin 10-15 min before release of aortic cross-clamp. The gradient between heat-exchanger and nasopharynx during rewarming will be maintained at 3oC. The rewarming will be stopped at 36,5oC
  Arms: Hypothermic CPB

SUMMARY:
Cardiopulmonary bypass (CPB) has been used successfully for cardiac surgery for over half a century. Hypothermia became a ubiquitous practice for adult patients undergoing CPB. To date, most studies have been conducted in coronary artery bypass graft (CABG) patients with conflicting results. Current evidence does not support one temperature management strategy for all patients. The purpose of this study is to compare the efficiency and safety of normothermic versus hypothermic CPB in valvular surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Isolated heart valve surgery
* Heart valve surgery plus CABG
* Age 20-80

Exclusion Criteria:

* urgent operation
* Left ventricle ejection fraction < 35%
* Decompensated congestive heart failure
* Chronic renal failure (glomerular filtration rate < 60 ml/min)
* Severe hepatic and pulmonary disease
* Bleeding diathesis or history of coagulopathy
* Planed deep hypothermic circulatory arrest
* History of acute myocardial infarction in the last 3 month
* Preoperative core temperature >37oC

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cardiac Troponin I release | 48 hours

SECONDARY OUTCOMES:
Need for Inotropic Support | First 48 postoperative hours
Rate of Perioperative Myocardial Infarction | First 48 postoperative hours
Rate of Type I and Type II neurological injury | 7 postoperative days
Rate of Dialysis-dependent acute renal failure | 7 postoperative days
Rate of infectious complications | 30 postoperative days
Total units of Red Blood Cells transfused | 7 postoperative days
Intensive Care Unit length of stay | 30 postoperative days
Hospital length of stay | 30 postoperative days
Rate of In-hospital mortality | 30 postoperative days
NT-proBNP release | First 24 postoperative hours
Bleeding from chest tubes | First 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Lomivorotov, MD, PhD, Principal Investigator — Research Institute of Pathology of Circulation
Locations (1):
- State Research Institute of Circulation Patholody, Novosibirsk, Russia

REFERENCES:
- [Result] Lomivorotov VV, Shmirev VA, Efremov SM, Ponomarev DN, Moroz GB, Shahin DG, Kornilov IA, Shilova AN, Lomivorotov VN, Karaskov AM. Hypothermic versus normothermic cardiopulmonary bypass in patients with valvular heart disease. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):295-300. doi: 10.1053/j.jvca.2013.03.009. Epub 2013 Aug 17. PMID 23962460